CLINICAL TRIAL: NCT01388348
Title: Diagnosis of Bladder Outlet Obstruction Using Dynamic Urine Vibration "Holter" in Comparison to Pressure Flow Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Ilan Leibovitch MD, Meir medical center
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: mmc 022-2011
Record Dates: First submitted 2011-02-15; First posted 2011-07-06 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2011-07

CONDITIONS: Bladder Outlet Obstruction
Keywords: benign prostatic hyperplasia (BPH); acoustic vibration
MeSH Terms: conditions — Urinary Bladder Neck Obstruction; Prostatic Hyperplasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dynamic Urine Vibration "Holter" (Experimental): each subject will undergo intervention for the diagnosis of bladder outlet obstruction first using the Dynamic Urine Vibration "Holter" and then urodynamically by pressure flow study
  Interventions: Device: Dynamic Urine Vibration "Holter"

INTERVENTIONS:
Device: Dynamic Urine Vibration "Holter" — each subject will undergo intervention for the diagnosis of bladder outlet obstruction first using the Dynamic Urine Vibration "Holter" and then urodynamically by pressure flow study

SUMMARY:
Current gold standard of bladder outlet diagnosis is pressure flow study. This study is invasive time consuming and requires expensive and complex set-up. In this study the investigators plan to evaluate an alternative technology that presumably is able to diagnose bladder outlet obstruction using a Dynamic Urine Vibration "Holter" based on a Urine Flow Vibration Analysis technology. The acoustic vibration sensor is a small device that records the vibration due to urine flow. The patient attaches the sensor to the penis using a disposable sensor patch for the duration of approximately one minute during one urination. The analysis is performed off-line and the results are compared to the results of a standard pressure flow study. The innovative technology for the diagnosis of bladder outlet obstruction is noninvasive, rapid and does not involve complex setup.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of benign prostatic hyperplasia (BPH)
* has indication for urodynamic evaluation

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-07; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Holter to confirm or exclude of bladder outlet obstruction | one recording at the time of urodynamic testing.approximatly one minute

CONTACTS AND LOCATIONS:
Locations (1):
- Meir Medical Center, Kfar Saba, Israel